CLINICAL TRIAL: NCT07107412
Title: Turkish Validity and Reliability of The General Rehabilitation Adherence Scale in Osteoarthritis Patients
Brief Title: Turkish General Rehabilitation Adherence Scale in Osteoarthritis Patients
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Hasan Gerçek, Lecturer, KTO Karatay University
Other Study IDs: KaratayUH15
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Translating the Questionnaire into Turkish and Related Processes — The first step is the translation from the original language to the other language. The ideal target in the translation phase is to use people who are familiar with the structure of the original language and who are familiar with the language. Two forward translation and one reverse translation methods will be applied after obtaining the written permission of the authors. After the completion of this phase, the terminological differences arising from the translators in the translation process from the original language to Turkish will be collected and discussed on the questions. The cultural adaptation study will be terminated by determining the equivalence between the Turkish version of the index and the English original. The final version of the questionnaire and the necessary changes will be arranged specific to the investigator's society and the authors of the original questionnaire will be consulted and the questionnaire will be finalized.
  Other: Validity The scale will be applied

SUMMARY:
Investigation of the Turkish Validity and Reliability of The General Rehabilitation Adherence Scale in Osteoarthritis Patients

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with osteoarthritis
* To be receiving physiotherapy
* Age between 18-85

Exclusion Criteria:

* Patients who do not want to participate
* Patients who filled out the questionnaire incompletely

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Validity | Baseline
  The scale will be applied by face-to-face technique and convergent (moderate-high correlation with optimism measure) and distant (low correlation with depression and anxiety measures) validity will be evaluated.
Reliability | Baseline
  The reliability of the materials will be tested with Cronbach alpha.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided